CLINICAL TRIAL: NCT03264495
Title: Recording Food Consumption in Patients Hospitalised in a Geriatric Centre
Brief Title: Measuring the Quantities of Food Consumed by Patients Hospitalised in a Geriatric Centre
Acronym: PESALI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: VAN WYMELBEKE 2016
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Age ≥ 65 Years; Hospitalisation in the Champmaillot Geriatric Centre

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Weight the food served minus the left-overs

SUMMARY:
The objective of the study is to measure the quantities of food consumed at each meal by a representative part of the population of patients hospitalised in each department of the Champmaillot Geriatric Centre.

To do so, the quantity eaten will be quantified by weighing the amounts served and subtracting the weight of the left-overs. These measurements will allow us to provide more appropriate meals in the second step.

ELIGIBILITY:
Inclusion Criteria:

* Persons aged ≥ 65 years
* Persons hospitalised in the Champmaillot Geriatric Centre

Exclusion Criteria:

* Persons at the end of life

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Elderly persons hospitalised at the Champmaillot Geriatric Centre
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Weigh the food served and the left-overs | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France